CLINICAL TRIAL: NCT05748899
Title: Effect of Applying Ujjayi Pranayama on Cortisol in Lupus Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdelhalim Elfahl, lecturer of physical therapy for Internal Medicine and Geriatrics, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004288
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): Group number 1 will receive home-based daily ujjayi pranayama for six weeks (fifteen minutes in the morning and 15 min in the evening, this training will be online supervised).
  Interventions: Behavioral: Ujjayi pranayama
- group number 2 (No Intervention): The group number 2 will not receive pranayama training, so it serves as control lupus group

INTERVENTIONS:
Behavioral: Ujjayi pranayama — this group will receive home-based daily ujjayi pranayama for six weeks (fifteen minutes in the morning and 15 min in the evening, this training will be online supervised).
  Arms: group number 1

SUMMARY:
stress vulnerability is very common in lupus patients, specifically women, hence the rates of depression , insomnia, easy fatigue perception, anxiety are high in those women. pranayama is a yogic intervention that may treat the above problems

DETAILED DESCRIPTION:
lupus patients, specifically 40 women, will divided to group number 1 and group number 2. the women in every group will be 20 women. Group number 1 will receive home-based ujjayi pranayama for six weeks (fifteen minutes in the morning and 15 min in the evening, this training will be online supervised). The group number 2 will not receive Ujjayi pranayama, so it serves as control lupus group

ELIGIBILITY:
Inclusion Criteria:

* 40 lupus women

Exclusion Criteria:

* lupus co-morbidities
* illiteracy

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity
Enrollment: 40 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
serum cortisol | it will be measured after 6 weeks
  it will be taken from women at morning

SECONDARY OUTCOMES:
systolic blood pressure | it will be measured after 6 weeks
  it will be assessed by manual sphygmomanometer
diastolic blood pressure | it will be measured after 6 weeks
  it will be assessed by manual sphygmomanometer
pulse rate | it will be measured after 6 weeks
  it is number of heart pulsation in minute
respiratory rate | it will be measured after 6 weeks
  it is number of respiration in minute
Pittsburgh Sleep Quality Index | it will be measured after 6 weeks
  it is a questionnaire assessing sleeping quality
Fatigue severity scale | it will be measured after 6 weeks
  it is a questionnaire assessing fatigue severity
Beck Depression Inventory | it will be measured after 6 weeks
  it is a questionnaire assessing depression
State Trait Anxiety Inventory | it will be measured after 6 weeks
  it is a questionnaire assessing Trait Anxiety
Stress Vulnerability Scale | it will be measured after 6 weeks
  it is a questionnaire assessing Stress Vulnerability

CONTACTS AND LOCATIONS:
Overall Officials: ahmed elfahl, Principal Investigator — Badr University
Locations (1):
- Badr University, Cairo, Egypt